CLINICAL TRIAL: NCT06536699
Title: A Randomised Non Inferiority Trial to Compare the Average Global Quality of Life Score Following Hypofractionated Radiotherapy Versus Conventional Fractionation in Head and Neck Cancers
Brief Title: Trial Comparing Avg. Global Qual of Lifescore in Hypo Frac. RT vs Conv. Frac. in H&N Cancers
Acronym: HYPORT-HN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/TMC/307/IRB11
Record Dates: First submitted 2024-07-01; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Radiation Treatment
Keywords: Hypofractionated radiotherapy; Head and Neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Intervention Model Description: Comparison of a shorter course of radiotherapy in 4 weeks with standard treatment of 6 weeks for head and neck cancers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy - conventional (Active Comparator): Conventional Radiotherapy of 66 Gy in 30 fractions in definitive setting and 60 Gy in 30 fractions in adjuvant setting Total Duration- 6 weeks
  Interventions: Radiation: Radiotherapy - Conventional
- Radiotherapy - hypofractionated (Experimental): Hypofractionated Radiotherapy of 55 Gy in 20 fractions in definitive setting and 52.5 Gy in 20 fractions in adjuvant setting. Total duration - 4 Weeks
  Interventions: Radiation: Radiotherapy - hypofractionated

INTERVENTIONS:
Radiation: Radiotherapy - hypofractionated — Hypofractionated Radiotherapy of 55 Gy in 20 fractions in definitive setting and 52.5 Gy in 20 fractions in adjuvant setting. Total duration - 4 Weeks
  Arms: Radiotherapy - hypofractionated
Radiation: Radiotherapy - Conventional — Conventional Radiotherapy of 66 Gy in 30 fractions in definitive setting and 60 Gy in 30 fractions in adjuvant setting. Total duration - 6 Weeks
  Arms: Radiotherapy - conventional

SUMMARY:
Radiotherapy forms an integral part of Head and Neck cancer treatment in both definitive as well as adjuvant setting. This study explores the use of hypofractionated radiotherapy, delivering 55Gy in 20 fractions over 4 weeks in comparison to the conventional approach which involves 70 Gy over 6 weeks.

Hypofractionated radiotherapy would result in significant benefits in terms of shortening the overall treatment time, countering accelerated hypofraction effects that typically arise after the 4th week. The new approach is also anticipated to offer resource and financial advantages, involving less machine time per patient, and potentially leading to better patient compliance. Previous studies on hypofractionation in Head and Neck cancer have demonstrated good local control and acceptable toxicity levels compared to conventional methods.

The primary objective of this study is to compare the average global quality of life following hypofractionated radiotherapy versus conventional fractionation, with secondary objectives including a comparison of locoregional control at 2 years and assessment of acute and late toxicities.

The study will require 600 eligible patients randomly assigned to either the hypofractionated or conventional arm. For definitive chemoradiation, the control arm will receive 66Gy in 30 fractions over 6 weeks, while the experimental arm will receive 55Gy in 20 fractions over 4 weeks, along with Inj Cisplatin @ 100mg/m2 3 weekly for 2 cycles. In the adjuvant setting control arm will receive 60Gy in 30 fractions over 6 weeks and experimental arm will receive 52.5Gy in 20 fractions over 4 weeks along with Inj Cisplatin @ 100mg /m2 3 weekly for 2 cycles for both arms based on histopathological indications.

Physician reported and patient reported acute toxicities like mucositis, dermatitis and dysphagia, weight loss, requirement and duration of feeding tubes as well as patients reported outcomes in the form of EORTC QLQ C30, HN43 and XeQoLS will be recorded both during and after treatment at regular intervals for 2 years.

The study's duration is five years, aiming to determine whether the hypofractionated schedule is non-inferior to conventional radiotherapy in terms of safety and disease-related outcomes

DETAILED DESCRIPTION:
Head and neck cancers comprise of cancers of arising from the epithelial lining of the lip, oral cavity, pharynx and larynx. The overall incidence of Head and Neck cancers continues to increase, despite decrease in the incidence of smoking suggestive of potential change in etiology. Presently Head and Neck cancer form the seventh most common cancer globally The primary treatment of oral cavity cancer comprises of surgery with adjuvant radiation with or without chemotherapy for locally advanced cancers or early-stage cancer in presence of high-risk factor. Cancers of the oropharynx are treated primarily with radiotherapy for early stage and chemoradiation for locally advanced disease. Laryngeal cancers are treated with either radiotherapy alone or chemoradiation, with surgery reserved for patients with laryngeal cartilage involvement or non-functional larynx.

Radiotherapy for head and neck cancer is delivered with conventional fractionation at 2- 2.2Gy per fraction to a total of 70 Gy dose equivalent. There are certain other altered fractionation types which has been tested like hyperfractionation with an intention to reduce late toxicities as well as accelerated and hypofractionation to counteract the effects of accelerated repopulation. Altered fractionation trials with hyperfractionation show increase in overall survival benefit when compared to radiotherapy alone but worse OS outcomes when compared to chemoradiation with lower toxicities. The advent of the COVID 19 pandemic popularised hypofractionated regimens with the ASTRO-ESTRO consensus statement which achieved a strong consensus about hypofractionated RT.

The addition of concurrent chemotherapy has been found to be superior compared to radiation alone in terms of locoregional control as well as overall survival. The MACH-NC meta analysis showed a 6.5% difference at 5 years and 3.6% at 10 years in favour of concurrent chemotherapy. The optimal dose of chemotherapy remains an important question. Although several studies have shown a significant improvement in overall survival with increasing cumulative cisplatin doses there might not be additional benefit of increasing dose of chemotherapy beyond a cumulative dose of 200mg/m2.

Through this study, the investigators aim to assess and compare the disease related outcomes, acute and late toxicities as well as the quality of life parameters of patients treated with hypofractionated radiotherapy along with two cycles 3 weekly concurrent chemotherapy versus those following the conventional chemotherapy regimen.

Rationale of study

1. Reduction in overall treatment time Squamous cell cancer of the Head and Neck region are rapidly proliferating cancers. Earlier studies have estimated a median value of labeling S-phase fraction (LI), duration, and estimated potential doubling time (Tpot) as 9%, 9 hours, and 5 days respectively. Although some studies failed to show any predictive value of pretreatment potential doubling time and labeling index in patients treated with conventional fractionation the effect of accelerated repopulation which is estimated to be triggered around about 4 +/- 1 weeks cannot be undermined. Several studies have shown a strong negative relation between overall treatment time and locoregional control and overall survival with an average loss of LRC from 1-1.2% per day to 12-14% per week. The dose time factor, also known as the K factor (or λ/α factor as used in some publications) ranges between 0.5 and 0.99 Gy/day with a recent meta-analysis on laryngeal cancers estimating it as 0.6 - 0.8.
2. Resource and financial benefits for patients, caregivers and hospitals. Reduction in total number of fractions will lead to an overall shorter duration of treatment and lesser number of hospital visits. For patients, an earlier end to treatment and lesser number of hospital visits will be a source of physical and financial relief. For caregivers, this will allow an earlier return to work or other responsibilities. For the healthcare system, it allows more patients to be offered treatment using the same resources.
3. Better patient compliance Reduced treatment time will increase patient compliance especially for patients who are taking treatment away from home.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. ECOG performance status 0 - 2.
3. Patients diagnosed with invasive squamous cell cancer of the head and neck region which includes lip, oral cavity, nasopharynx, oropharynx, hypopharynx, supraglottis, glottis and subglottis.
4. Patients who are being treated with curative intent treatment either with surgery followed by adjuvant radiotherapy with or without chemotherapy or definitive chemoradiation.
5. Patients must have a histopathological proof of malignancy, such as biopsy or post operative histopathology report. Biopsies or surgeries done outside must have been reviewed for pathological confirmation and specimen adequacy at the treating institute.
6. Patients with non metastatic cancer, optimally staged with the following:

   1. Contrast enhanced CT scan of the neck and thorax for cancer lip, oral cavity, oropharynx, hypopharynx, supraglottis, glottis and subglottis
   2. Magnetic Resonance Imaging of the neck and CT thorax for cancer of nasopharynx

Exclusion Criteria:

1. Concurrent illness like severe cardiac, renal or hepatic dysfunction and, including severe infection that may jeopardise the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety
2. Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-08-07 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
To compare the average global quality of life score following hypofractionated radiotherapy versus conventional fractionation in head and neck cancer | 2 Years
  Patients reported outcomes in the form of EORTC QLQ C30 questionnaire at regular designated intervals using electronic patient reported outcome monitoring systems (e-PROMS).
  EORTC QLQ C30 stands for European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire C30.
  The score will range from 0 to 100 as per the Scoring of the EORTC QLQ-C30 version 3.0.
  A higher score will denote a better quality of life.

SECONDARY OUTCOMES:
To compare the locoregional control at 2 years between the hypofractionated and conventional arm. | 2 Years
  To get a Radiological assessment done 3 months post treatment and then followup the patient clinically and only get a radiological correlation if suggested clinically.
To compare acute and late toxicities of hypofractionated radiotherapy with conventional fractionation | 2 Years
  To compare physician reported and patient reported acute toxicities like mucositis, dermatitis and dysphagia between the two groups using weekly assessment of acute toxicities using the RTOG and CTCAE v5 criteria during radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjoy Sanjoy, MRCP,FRCR, Principal Investigator — Tata Medical Center
Locations (1):
- Tata Medical Center, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identiﬁcation (text, tables, ﬁgures, and appendices).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Baujat B, Bourhis J, Blanchard P, Overgaard J, Ang KK, Saunders M, Le Maitre A, Bernier J, Horiot JC, Maillard E, Pajak TF, Poulsen MG, Bourredjem A, O'Sullivan B, Dobrowsky W, Andrzej H, Skladowski K, Hay JH, Pinto LH, Fu KK, Fallai C, Sylvester R, Pignon JP; MARCH Collaborative Group. Hyperfractionated or accelerated radiotherapy for head and neck cancer. Cochrane Database Syst Rev. 2010 Dec 8;2010(12):CD002026. doi: 10.1002/14651858.CD002026.pub2. PMID 21154350
- [Background] Bentzen SM, Rosenblatt E, Gupta T, Agarwal JP, Laskar SG, Bhasker S, et al. Randomized Controlled Trial of Hypofractionated vs. Normo-fractionated Accelerated Radiation Therapy with or without Cisplatin for Locally Advanced Head and Neck Squamous Cell Carcinoma (HYPNO). International Journal of Radiation Oncology*Biology*Physics. 2023 Nov;117(4):e2
- [Background] Fu KK, Pajak TF, Trotti A, Jones CU, Spencer SA, Phillips TL, Garden AS, Ridge JA, Cooper JS, Ang KK. A Radiation Therapy Oncology Group (RTOG) phase III randomized study to compare hyperfractionation and two variants of accelerated fractionation to standard fractionation radiotherapy for head and neck squamous cell carcinomas: first report of RTOG 9003. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):7-16. doi: 10.1016/s0360-3016(00)00663-5. PMID 10924966
- [Background] Thomson DJ, Palma D, Guckenberger M, Balermpas P, Beitler JJ, Blanchard P, Brizel D, Budach W, Caudell J, Corry J, Corvo R, Evans M, Garden AS, Giralt J, Gregoire V, Harari PM, Harrington K, Hitchcock YJ, Johansen J, Kaanders J, Koyfman S, Langendijk JA, Le QT, Lee N, Margalit D, Mierzwa M, Porceddu S, Soong YL, Sun Y, Thariat J, Waldron J, Yom SS. Practice recommendations for risk-adapted head and neck cancer radiotherapy during the COVID-19 pandemic: An ASTRO-ESTRO consensus statement. Radiother Oncol. 2020 Oct;151:314-321. doi: 10.1016/j.radonc.2020.04.019. Epub 2020 Jul 27. PMID 32730830
- [Background] Gupta T, Ghosh-Laskar S, Agarwal JP. Resource-sparing curative-intent hypofractionated-accelerated radiotherapy in head and neck cancer: More relevant than ever before in the COVID era. Oral Oncol. 2020 Dec;111:105045. doi: 10.1016/j.oraloncology.2020.105045. Epub 2020 Oct 20. PMID 33091846
- [Background] Adelstein DJ, Li Y, Adams GL, Wagner H Jr, Kish JA, Ensley JF, Schuller DE, Forastiere AA. An intergroup phase III comparison of standard radiation therapy and two schedules of concurrent chemoradiotherapy in patients with unresectable squamous cell head and neck cancer. J Clin Oncol. 2003 Jan 1;21(1):92-8. doi: 10.1200/JCO.2003.01.008. PMID 12506176
- [Background] Forastiere AA, Goepfert H, Maor M, Pajak TF, Weber R, Morrison W, Glisson B, Trotti A, Ridge JA, Chao C, Peters G, Lee DJ, Leaf A, Ensley J, Cooper J. Concurrent chemotherapy and radiotherapy for organ preservation in advanced laryngeal cancer. N Engl J Med. 2003 Nov 27;349(22):2091-8. doi: 10.1056/NEJMoa031317. PMID 14645636
- [Background] Cooper JS, Pajak TF, Forastiere AA, Jacobs J, Campbell BH, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Machtay M, Ensley JF, Chao KS, Schultz CJ, Lee N, Fu KK; Radiation Therapy Oncology Group 9501/Intergroup. Postoperative concurrent radiotherapy and chemotherapy for high-risk squamous-cell carcinoma of the head and neck. N Engl J Med. 2004 May 6;350(19):1937-44. doi: 10.1056/NEJMoa032646. PMID 15128893
- [Background] Bernier J, Domenge C, Ozsahin M, Matuszewska K, Lefebvre JL, Greiner RH, Giralt J, Maingon P, Rolland F, Bolla M, Cognetti F, Bourhis J, Kirkpatrick A, van Glabbeke M; European Organization for Research and Treatment of Cancer Trial 22931. Postoperative irradiation with or without concomitant chemotherapy for locally advanced head and neck cancer. N Engl J Med. 2004 May 6;350(19):1945-52. doi: 10.1056/NEJMoa032641. PMID 15128894
- [Background] Lacas B, Carmel A, Landais C, Wong SJ, Licitra L, Tobias JS, Burtness B, Ghi MG, Cohen EEW, Grau C, Wolf G, Hitt R, Corvo R, Budach V, Kumar S, Laskar SG, Mazeron JJ, Zhong LP, Dobrowsky W, Ghadjar P, Fallai C, Zakotnik B, Sharma A, Bensadoun RJ, Ruo Redda MG, Racadot S, Fountzilas G, Brizel D, Rovea P, Argiris A, Nagy ZT, Lee JW, Fortpied C, Harris J, Bourhis J, Auperin A, Blanchard P, Pignon JP; MACH-NC Collaborative Group. Meta-analysis of chemotherapy in head and neck cancer (MACH-NC): An update on 107 randomized trials and 19,805 patients, on behalf of MACH-NC Group. Radiother Oncol. 2021 Mar;156:281-293. doi: 10.1016/j.radonc.2021.01.013. Epub 2021 Jan 27. PMID 33515668
- [Background] Haselow RE, Warshaw MG, Oken MM, et al. Radiation alone versus radiation with weekly low dose cis-platinum in unresectable cancer of the head and neck. In: Fee WE Jr, Goepfert H, Johns ME, et al, editors. Head and Neck Cancer, vol. II. Toronto, Canada and Philadelphia, PA: BC Decker; 1990. pp 279-281.
- [Background] Quon H, Leong T, Haselow R, Leipzig B, Cooper J, Forastiere A. Phase III study of radiation therapy with or without cis-platinum in patients with unresectable squamous or undifferentiated carcinoma of the head and neck: an intergroup trial of the Eastern Cooperative Oncology Group (E2382). Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):719-25. doi: 10.1016/j.ijrobp.2010.06.038. Epub 2010 Oct 1. PMID 20888709
- [Background] Jeremic B, Shibamoto Y, Stanisavljevic B, Milojevic L, Milicic B, Nikolic N. Radiation therapy alone or with concurrent low-dose daily either cisplatin or carboplatin in locally advanced unresectable squamous cell carcinoma of the head and neck: a prospective randomized trial. Radiother Oncol. 1997 Apr;43(1):29-37. doi: 10.1016/s0167-8140(97)00048-0. PMID 9165134
- [Background] Jeremic B, Milicic B, Dagovic A, Vaskovic Z, Tadic L. Radiation therapy with or without concurrent low-dose daily chemotherapy in locally advanced, nonmetastatic squamous cell carcinoma of the head and neck. J Clin Oncol. 2004 Sep 1;22(17):3540-8. doi: 10.1200/JCO.2004.10.076. PMID 15337803
- [Background] Jeremic B, Shibamoto Y, Milicic B, Nikolic N, Dagovic A, Aleksandrovic J, Vaskovic Z, Tadic L. Hyperfractionated radiation therapy with or without concurrent low-dose daily cisplatin in locally advanced squamous cell carcinoma of the head and neck: a prospective randomized trial. J Clin Oncol. 2000 Apr;18(7):1458-64. doi: 10.1200/JCO.2000.18.7.1458. PMID 10735893
- [Background] Huguenin P, Beer KT, Allal A, Rufibach K, Friedli C, Davis JB, Pestalozzi B, Schmid S, Thoni A, Ozsahin M, Bernier J, Topfer M, Kann R, Meier UR, Thum P, Bieri S, Notter M, Lombriser N, Glanzmann C. Concomitant cisplatin significantly improves locoregional control in advanced head and neck cancers treated with hyperfractionated radiotherapy. J Clin Oncol. 2004 Dec 1;22(23):4665-73. doi: 10.1200/JCO.2004.12.193. Epub 2004 Nov 8. PMID 15534360
- [Background] Ghadjar P, Simcock M, Studer G, Allal AS, Ozsahin M, Bernier J, Topfer M, Zimmermann F, Betz M, Glanzmann C, Aebersold DM; Swiss Group for Clinical Cancer Research (SAKK). Concomitant cisplatin and hyperfractionated radiotherapy in locally advanced head and neck cancer: 10-year follow-up of a randomized phase III trial (SAKK 10/94). Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):524-31. doi: 10.1016/j.ijrobp.2010.11.067. Epub 2011 Feb 16. PMID 21300466
- [Background] Fountzilas G, Ciuleanu E, Dafni U, Plataniotis G, Kalogera-Fountzila A, Samantas E, Athanassiou E, Tzitzikas J, Ciuleanu T, Nikolaou A, Pantelakos P, Zaraboukas T, Zamboglou N, Daniilidis J, Ghilezan N. Concomitant radiochemotherapy vs radiotherapy alone in patients with head and neck cancer: a Hellenic Cooperative Oncology Group Phase III Study. Med Oncol. 2004;21(2):95-107. doi: 10.1385/MO:21:2:095. PMID 15299181
- [Background] Sharma A, Mohanti BK, Thakar A, Bahadur S, Bhasker S. Concomitant chemoradiation versus radical radiotherapy in advanced squamous cell carcinoma of oropharynx and nasopharynx using weekly cisplatin: a phase II randomized trial. Ann Oncol. 2010 Nov;21(11):2272-2277. doi: 10.1093/annonc/mdq219. Epub 2010 Apr 28. PMID 20427350
- [Background] Strojan P, Vermorken JB, Beitler JJ, Saba NF, Haigentz M Jr, Bossi P, Worden FP, Langendijk JA, Eisbruch A, Mendenhall WM, Lee AW, Harrison LB, Bradford CR, Smee R, Silver CE, Rinaldo A, Ferlito A. Cumulative cisplatin dose in concurrent chemoradiotherapy for head and neck cancer: A systematic review. Head Neck. 2016 Apr;38 Suppl 1:E2151-8. doi: 10.1002/hed.24026. Epub 2015 Jul 14. PMID 25735803
- [Background] Ang K, Zhang Q, Wheeler RH, et al. A phase III trial (RTOG 0129) of two radiation-cisplatin regimens for head and neck carcinomas (HNC): impact of radiation and cisplatin intensity on outcome. J Clin Oncol 2010; 28(suppl):abstract 5507.
- [Background] Lee AW, Tung SY, Ngan RK, Chappell R, Chua DT, Lu TX, Siu L, Tan T, Chan LK, Ng WT, Leung TW, Fu YT, Au GK, Zhao C, O'Sullivan B, Tan EH, Lau WH. Factors contributing to the efficacy of concurrent-adjuvant chemotherapy for locoregionally advanced nasopharyngeal carcinoma: combined analyses of NPC-9901 and NPC-9902 Trials. Eur J Cancer. 2011 Mar;47(5):656-66. doi: 10.1016/j.ejca.2010.10.026. Epub 2010 Nov 26. PMID 21112774
- [Background] Corvo R, Giaretti W, Sanguineti G, Geido E, Orecchia R, Barra S, Margarino G, Bacigalupo A, Vitale V. Potential doubling time in head and neck tumors treated by primary radiotherapy: preliminary evidence for a prognostic significance in local control. Int J Radiat Oncol Biol Phys. 1993 Dec 1;27(5):1165-72. doi: 10.1016/0360-3016(93)90539-8. PMID 8262843
- [Background] Awwad HK, Lotayef M, Shouman T, Begg AC, Wilson G, Bentzen SM, Abd El-Moneim H, Eissa S. Accelerated hyperfractionation (AHF) compared to conventional fractionation (CF) in the postoperative radiotherapy of locally advanced head and neck cancer: influence of proliferation. Br J Cancer. 2002 Feb 12;86(4):517-23. doi: 10.1038/sj.bjc.6600119. PMID 11870530
- [Background] Gonzalez Ferreira JA, Jaen Olasolo J, Azinovic I, Jeremic B. Effect of radiotherapy delay in overall treatment time on local control and survival in head and neck cancer: Review of the literature. Rep Pract Oncol Radiother. 2015 Sep-Oct;20(5):328-39. doi: 10.1016/j.rpor.2015.05.010. Epub 2015 Jul 4. PMID 26549990
- [Background] Dale RG, Hendry JH, Jones B, Robertson AG, Deehan C, Sinclair JA. Practical methods for compensating for missed treatment days in radiotherapy, with particular reference to head and neck schedules. Clin Oncol (R Coll Radiol). 2002 Oct;14(5):382-93. doi: 10.1053/clon.2002.0111. PMID 12555877
- [Background] Goswami U, Banerjee S, Dutta S, Bera A. TREATMENT OUTCOME AND TOXICITY OF HYPOFRACTIONATED RADIOTHERAPY WITH CONCOMITANT CHEMOTHERAPY VERSUS CONVENTIONAL FRACTIONATED CONCOMITANT CHEMORADIATION IN LOCALLY ADVANCED HEAD-AND-NECK CARCINOMA: A COMPARATIVE STUDY. Asian J Pharm Clin Res. 2022 Jul 7;167-71.
- [Background] Sanghera P, McConkey C, Ho KF, Glaholm J, Hartley A. Hypofractionated accelerated radiotherapy with concurrent chemotherapy for locally advanced squamous cell carcinoma of the head and neck. Int J Radiat Oncol Biol Phys. 2007 Apr 1;67(5):1342-51. doi: 10.1016/j.ijrobp.2006.11.015. Epub 2007 Jan 22. PMID 17241752
- [Background] Jegannathen A, Mais K, Sykes A, Lee L, Yap B, Birzgalis A, Homer J, Ryder WD, Slevin N. Synchronous chemoradiotherapy in patients with locally advanced squamous cell carcinoma of the head and neck using capecitabine: a single-centre, open-label, single-group phase II study. Clin Oncol (R Coll Radiol). 2011 Mar;23(2):149-58. doi: 10.1016/j.clon.2010.09.010. Epub 2010 Oct 14. PMID 20951012
- [Background] Chan AK, Sanghera P, Choo BA, McConkey C, Mehanna H, Parmar S, Pracy P, Glaholm J, Hartley A. Hypofractionated accelerated radiotherapy with concurrent carboplatin for locally advanced squamous cell carcinoma of the head and neck. Clin Oncol (R Coll Radiol). 2011 Feb;23(1):34-9. doi: 10.1016/j.clon.2010.07.015. Epub 2010 Sep 21. PMID 20863676
- [Background] Benghiat H., Sanghera P., Cashmore J. Four-week hypofractionated accelerated intensity modulated radiotherapy and synchronous carboplatin or cetuximab in biologically staged oropharyngeal carcinoma. Cancer Clin Oncol. 2014;3(2):2.
- [Background] Jacinto AA, Batalha Filho ES, Viana LS, De Marchi P, Capuzzo RC, Gama RR, Boldrini Junior D, Santos CR, Pinto GDJ, Dias JM, Canton HP, Carvalho R, Radicchi LA, Bentzen S, Zubizarreta E, Carvalho AL. Feasibility of concomitant cisplatin with hypofractionated radiotherapy for locally advanced head and neck squamous cell carcinoma. BMC Cancer. 2018 Oct 23;18(1):1026. doi: 10.1186/s12885-018-4893-5. PMID 30352576
- [Background] Mayo ZS, Ilori EO, Matia B, Smile TD, Fleming CW, Reddy CA, Scharpf J, Lamarre ED, Prendes BL, Ku J, Burkey BB, Joshi NP, Woody NM, Koyfman SA, Campbell SR. Limited Toxicity of Hypofractionated Intensity Modulated Radiation Therapy for Head and Neck Cancer. Anticancer Res. 2022 Apr;42(4):1845-1849. doi: 10.21873/anticanres.15660. PMID 35347002
- [Background] Piras A, Boldrini L, Menna S, Venuti V, Pernice G, Franzese C, Angileri T, Daidone A. Hypofractionated Radiotherapy in Head and Neck Cancer Elderly Patients: A Feasibility and Safety Systematic Review for the Clinician. Front Oncol. 2021 Nov 12;11:761393. doi: 10.3389/fonc.2021.761393. eCollection 2021. PMID 34868976
- [Background] Musoro JZ, Coens C, Singer S, Tribius S, Oosting SF, Groenvold M, Simon C, Machiels JP, Gregoire V, Velikova G, Cocks K, Sprangers MAG, King MT, Bottomley A; EORTC Head and Neck and Quality of Life Groups. Minimally important differences for interpreting European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 scores in patients with head and neck cancer. Head Neck. 2020 Nov;42(11):3141-3152. doi: 10.1002/hed.26363. Epub 2020 Jul 6. PMID 32627261
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338